CLINICAL TRIAL: NCT04814654
Title: CHALO! 2.0: A Mobile Technology Based Intervention to Accelerate HIV Testing and Linkage to Preventive Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: The Humsafar Trust (Unknown); National Institute of Mental Health (NIMH) (NIH); Hunter College of City University of New York (Other); Fenway Community Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-9471; R01MH119001 (NIH)
Record Dates: First submitted 2021-03-15; First posted 2021-03-24 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Hiv
Keywords: HIV screening; HIV testing; HIV prevention; HIV linkage to care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Subjects meeting all eligibility criteria will be randomized to one of three study arms. Participants will be assigned either to CHALO! 2.0 (intervention), to an Attention-Matched Control, or to a Digital Coupon for free HIV testing only arm. After baseline survey completion, the research team will use random blocked design, with a fixed block size, to stratify randomization by prior HIV testing history (never tested vs. not tested in >6 months).
Who Masked: Participant, Investigator
Masking Description: The Data Manager (who has no contact with study participants) will assign participants to a study group and cross-reference encrypted files with our technology consultant. Participants will be unaware of arm assignment and will receive automated messages to complete online surveys. Study staff collecting HIV testing and linkage-to-care outcomes will also be blinded to the participants' study arm. Finally, the team of Virtual Peers will not be informed of study hypothesis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHALO! 2.0 (Experimental): MSM randomized to this arm will receive twice weekly digital media messages for 12 weeks about HIV, HIV-testing, prevention, and treatment and a a link to a study-specific webpage listing MSM specific testing, prevention, and care resources. Participants will also be able to interact with online outreach workers.
  Interventions: Behavioral: CHALO! 2.0
- Attention-matched control (AMC) (Active Comparator): MSM randomized to the AMC arm will receive twice weekly digital media messages for 12 weeks about general health and a link to a study-specific webpage listing testing resources and MSM-specific services. Participants will also be able to interact with online outreach workers.
  Interventions: Behavioral: Attention-matched control (AMC)
- Digital coupon only control (DCO) (Active Comparator): MSM randomized to the DCO arm will receive, at study entry, a digital coupon for free HIV testing and a study specific webpage link listing testing and MSM specific services.
  Interventions: Behavioral: Digital coupon only (DCO)

INTERVENTIONS:
Behavioral: CHALO! 2.0 — The components of the intervention are:
  Contents of digital-media (sent twice/week for 12 weeks) on the following topics: HIV testing, prevention, treatment, linkage-to-care; Personalized digital coupon for free testing; Webpage listing testing/ care sites; access to online outreach workers.
  Arms: CHALO! 2.0
Behavioral: Attention-matched control (AMC) — The components of the intervention are:
  Contents of digital-media (sent twice/week for 12 weeks) only related to general health information; Personalized digital coupon for free testing; Webpage listing testing/ care sites; access to online outreach workers.
  Arms: Attention-matched control (AMC)
Behavioral: Digital coupon only (DCO) — The components of the intervention are:
  Digital coupon for free HIV testing; Webpage listing testing/ care sites; access to online outreach workers.
  Arms: Digital coupon only control (DCO)

SUMMARY:
While HIV prevalence among Men Seeking Men (MSM) in India is 10-15 times higher than in the general population (4.3% vs 0.3%), current interventions for Indian MSM have limited reach. In order to reduce the burden of HIV in MSM, innovative, far-reaching prevention and treatment strategies are needed. Guided by the increase access to internet-based social and mobile technologies (SMT) (e.g., SMS, WhatsApp, dating apps) globally and in India, this is a 3-arm parallel, pragmatic randomized controlled trial of community-developed, theory based behavioral intervention (CHALO! 2.0) delivered via WhatsApp (secure SMS application) compared to an Attention-Matched Control, or a Digital Coupon for free HIV testing only control conditions. The primary outcomes are HIV-testing at 6 months (3 months after the end of the intervention) and linkage-to-preventive care (counseling or pre-exposure prophylaxis) at 12 months. The secondary outcomes are the frequency of HIV-testing by 18 months.

ELIGIBILITY:
Inclusion Criteria:

* live or work in Mumbai or Thane
* fluent in Hindi or English
* have had anal sex with men in the past one year
* report that they have either never been tested for HIV, are unaware of HIV test results, or are HIV-negative with last HIV test at any time, and have engaged in anal sex since last HIV test
* able to provide and verify a WhatsApp mobile number and email address
* willing to answer online surveys for 18 months

Exclusion Criteria:

* participating in a concurrent HIV-related study
* intention to move out of the Mumbai metropolitan area in the next six months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified cis-gendered men
Enrollment: 1004 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viraj V Patel, MD, MPH, Principal Investigator — Associate Professor, Division of General Internal Medicine, Albert Einstein College of Medicine
Locations (1):
- The Humsafar Trust, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
IPD results will not be publicly deposited. IPD will be available on appropriate request and IRB/ethics review board approval. An executed Data Use Agreement must accompany all requests for data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following study publication
Access Criteria: Data requestor must obtain an executed Data Use Agreement and IRB/ethics board approvals.

REFERENCES:
- [Derived] Chaudary J, Rawat S, Dange A, Golub SA, Kim RS, Chakrapani V, Mayer KH, Arnsten J, Patel VV. The CHALO! 2.0 mHealth-Based Multilevel Intervention to Promote HIV Testing and Linkage-to-Care Among Men Who Have Sex with Men in Mumbai, India: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Nov 5;13:e59873. doi: 10.2196/59873. PMID 39499921

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For this study a total of 1191 were consented. Upon quality checking 187 participants were excluded after enrollment. After these exclusions 1004 participants were considered enrolled and were randomized.
Groups:
- CHALO! 2.0: MSM randomized to this arm will receive twice weekly digital media messages for 12 weeks about HIV, HIV-testing, prevention, and treatment and a a link to a study-specific webpage listing MSM specific testing, prevention, and care resources. Participants will also be able to interact with online outreach workers.
  CHALO! 2.0: The components of the intervention are:
  Contents of digital-media (sent twice/week for 12 weeks) on the following topics: HIV testing, prevention, treatment, linkage-to-care; Personalized digital coupon for free testing; Webpage listing testing/ care sites; access to online outreach workers.
- Attention-matched Control (AMC): MSM randomized to the AMC arm will receive twice weekly digital media messages for 12 weeks about general health and a link to a study-specific webpage listing testing resources and MSM-specific services. Participants will also be able to interact with online outreach workers.
  Attention-matched control (AMC): The components of the intervention are:
  Contents of digital-media (sent twice/week for 12 weeks) only related to general health information; Personalized digital coupon for free testing; Webpage listing testing/ care sites; access to online outreach workers.
- Digital Coupon Only Control (DCO): MSM randomized to the DCO arm will receive, at study entry, a digital coupon for free HIV testing and a study specific webpage link listing testing and MSM specific services.
  Digital coupon only (DCO): The components of the intervention are:
  Digital coupon for free HIV testing; Webpage listing testing/ care sites; access to online outreach workers.
Period: Overall Study
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Started | 339 | 332 | 333
Completed | 169 | 165 | 176
Not Completed | 170 | 167 | 157
Not completed — due to administrative issues, implementation partner was unable to continue study activities. | 170 | 167 | 157

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO) | Total
Number analyzed (Participants) | 339 | 332 | 333 | 1004
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 339 | 332 | 333 | 1004
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28 (7) | 28 (7) | 28 (7) | 28 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 339 | 332 | 333 | 1004
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 339 | 332 | 333 | 1004

OUTCOME MEASURES:

1. Primary Outcome: Verified HIV Testing
Description: Verified HIV testing was assessed as a dichotomous measure (yes/no) of receipt of a documented HIV test. The number/percentage of participants who were verified to have been HIV tested within 6 months of randomization is summarized by study arm/group.
Time Frame: Within 6 months from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 339 | 332 | 333
Participants | 30 | 30 | 29
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.989, Chi-squared
Statistical Analysis 2: Comparison: CHALO! 2.0 vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.949, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.60 to 1.74]
Statistical Analysis 3: Comparison: Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.882, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.61 to 1.78]

2. Primary Outcome: Linkage to Prevention
Description: Linkage to prevention was assessed as a dichotomous (yes/no) measure and defined as a composite of either receipt of counseling or PrEP use within 12 months of randomization. The number/percentage of participants who meet the linkage to care composite criteria is summarized by study arm/group.
Time Frame: Within 12 months from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 339 | 332 | 333
Participants | 31 | 47 | 32
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = .0726, Chi-squared

3. Secondary Outcome: Frequency of HIV Testing
Description: Among participants who were tested, frequency of HIV testing is defined as the average (mean) number of verified HIV tests per participant within 18 months from randomization. Frequency of HIV testing is a measure of public health intervention effectiveness. Results are summarized by study arm/group using descriptive statistics.
Time Frame: Within 18 months from randomization
Population: This analysis is among the total of N=164 total who had a verified HIV test within 18 months of randomization.
Measure: Mean (Standard Deviation); unit: HIV tests per participant
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 57 | 63 | 44
HIV tests per participant | 1.77 (1.0) | 1.27 (0.6) | 1.78 (1.1)
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); 12 month timepoint; Test type: Superiority; p = 0.918, Kruskal-Wallis
Statistical Analysis 2: Comparison: CHALO! 2.0 vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.948, Kruskal-Wallis
Statistical Analysis 3: Comparison: Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = .0766, Kruskal-Wallis

4. Secondary Outcome: Receipt of a Verified HIV Test
Description: Receipt of a verified HIV test within 18 months of randomization was assessed as a dichotomous (yes/no) measure. The number/percentage of participants who were verified to have received HIV testing at each protocol-specified timepoint (i.e., within 12 months and within 18 months of randomization) is summarized by study arm/group.
Time Frame: Within 12 and 18 months from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 339 | 332 | 333
Participants
  12 months | 41 | 52 | 37
  18 months | 57 | 63 | 44
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); 12 months; Test type: Superiority; p = 0.1839, Chi-squared
Statistical Analysis 2: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); 18 months; Test type: Superiority; p = .127, Chi-squared

5. Secondary Outcome: Self-reported HIV Test
Description: Self-reported HIV test within 6 months of randomization was assessed as a dichotomous (yes/no) measure. The number/percentage of participants who self-reported as having been HIV tested, but were unverified, within 6 months from randomization is summarized by study arm/group.
Time Frame: Within 6 months from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 339 | 332 | 333
Participants | 119 | 107 | 113
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.7313, Chi-squared

6. Secondary Outcome: Linkage to HIV Treatment for HIV Positive Participants
Description: Linkage to HIV treatment was assessed as a dichotomous (yes/no) measure of whether participants who tested HIV-positive formally sought treatment. The number/percentage of HIV positive participants who sought treatment within 12 months from randomization is summarized by study arm/group.
Time Frame: Within 12 months from randomization
Population: This analysis is among people who tested positive and had a confirmed positive HIV test.
Measure: Count of Participants; unit: Participants
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 4 | 6 | 5
Participants | 3 | 6 | 5
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.1839, Chi-squared

7. Secondary Outcome: Linkage to Antiretroviral Therapy (ART) Initiation for HIV Positive Participants
Description: Linkage to ART initiation was assessed as a dichotomous (yes/no) measure of whether participants who tested HIV positive initiated ART treatment. The number/percentage of HIV positive participants who initiated ART within 12 months from randomization is summarized by study arm/group.
Time Frame: Within 12 months from randomization
Population: This analysis is among people who tested positive and had a confirmed positive HIV test.
Measure: Count of Participants; unit: Participants
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 4 | 6 | 5
Participants | 3 | 6 | 5
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.2667, Fisher Exact

8. Secondary Outcome: Linkage to Pre-Exposure Prophylaxis (PrEP) for HIV Negative Participants
Description: Linkage to PrEP was assessed as a dichotomous (yes/no) measure of whether participants who tested HIV negative were on a PrEP regimen. The number/percentage of HIV negative participants who were on a PrEP regimen within 12 months from randomization is summarized by study arm/group.
Time Frame: Within 12 months from randomization
Population: This outcome was only among individuals who tested HIV negative.
Measure: Count of Participants; unit: Participants
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 37 | 46 | 32
Participants | 1 | 1 | 0
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.999, Fisher Exact

9. Secondary Outcome: Linkage to Counseling
Description: Linkage to counseling was assessed as a dichotomous (yes/no) measure of whether participants received counseling treatment. The number/percentage of participants who received status neutral counseling treatment within 12 months from randomization is summarized by study arm/group.
Time Frame: Within 12 months from randomization
Population: Linkage to counselling is for all participants irrespective of whether participants were HIV positive or negative.
Measure: Count of Participants; unit: Participants
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 339 | 332 | 333
Participants | 50 | 59 | 41
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.1414, Chi-squared

10. Secondary Outcome: Sexual Behaviors - Consistent Condom Use
Description: Sexual Behavior will be evaluated based on consistent condom use. Specifically, this measure will be assessed as a dichotomous (yes/no) measure as to whether participants engaged in condomless anal sex during the study. Results will be summarized by study arm.
Time Frame: Within 18 months from randomization
Population: Analyzed among all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 339 | 332 | 333
Participants | 63 | 73 | 60
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.425, Chi-squared

11. Other Pre Specified Outcome: Linkage to Care
Description: a composite of linkage to PrEP, counseling, or HIV treatment (yes/no)
Time Frame: Within 18 months from randomization
Reporting Status: Not Posted

12. Other Pre Specified Outcome: PEP Use
Description: a dichotomous measure (yes/no) of whether a participant sought PEP treatment
Time Frame: within six months from randomization
Reporting Status: Not Posted

13. Other Pre Specified Outcome: HIV Testing
Description: a dichotomous measure (yes/no) of whether a participant intends to obtain an HIV test in the next one month
Time Frame: within six months from randomization
Reporting Status: Not Posted

14. Other Pre Specified Outcome: STI Testing / Treatment
Description: a dichotomous measure (yes/no) of whether a participant sought further STI testing or treatment
Time Frame: within six months from randomization
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Type of Site Accessed
Description: Type of prevention or treatment care site accessed (i.e., Humsafar Trust, public institution, private institution)
Time Frame: within six months from randomization
Reporting Status: Not Posted

16. Other Pre Specified Outcome: HIV and PrEP Knowledge
Description: The HIV and PrEP knowledge retained by participants
Time Frame: within six months from randomization
Reporting Status: Not Posted

17. Other Pre Specified Outcome: HIV and MSM Stigma
Description: Stigma related to HIV and men who have sex with men (MSM) reported by participants
Time Frame: within six months from randomization
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Risk Perception
Description: The risk perception reported by participants
Time Frame: within six months from randomization
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Self-efficacy
Description: The self-efficacy reported by participants
Time Frame: within six months from randomization
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Social Support
Description: The social support reported by participants
Time Frame: within six months from randomization
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Alcohol and Substance Use
Description: The alcohol and substance usage reported by participants
Time Frame: within six months from randomization
Reporting Status: Not Posted

22. Secondary Outcome: Sexual Behaviors - Number of Sexual Partners
Description: Sexual Behavior will be also be evaluated based on the number of sexual partners a participant had during the course of the study. This measure will be summarized by study arm using basic descriptive statistics.
Time Frame: Within 18 months from randomization
Population: Analyzed among all participants.
Measure: Median (Inter-Quartile Range); unit: sexual partners
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
Number analyzed (Participants) | 339 | 332 | 333
sexual partners | 3 [1 to 3] | 3 [1 to 3] | 2 [1 to 3]
Statistical Analysis 1: Comparison: CHALO! 2.0 vs Attention-matched Control (AMC) vs Digital Coupon Only Control (DCO); Test type: Superiority; p = 0.9183, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Approximately 18 months
Arm/Group | CHALO! 2.0 | Attention-matched Control (AMC) | Digital Coupon Only Control (DCO)
All-Cause Mortality (participants affected / at risk) | 0/339 | 0/332 | 0/333
Serious Adverse Events (participants affected / at risk) | 0/339 | 0/332 | 0/333
Other Adverse Events (participants affected / at risk) | 1/339 | 0/332 | 0/333
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CHALO! 2.0 (N=339) | Attention-matched Control (AMC) (N=332) | Digital Coupon Only Control (DCO) (N=333)
Emotional distress (Social circumstances) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04814654/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT04814654/ICF_000.pdf